CLINICAL TRIAL: NCT03851562
Title: Prospective, Unicentric, Randomized, Parallel, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate Intravenous Infusion of Prostaglandins as Therapy in Patients With Anterior Non-arteritic Ischemic Optic Neuropathy
Brief Title: Intravenous Infusion of Prostaglandins as Therapy in Patients With Anterior Non-arteritic Ischemic Optic Neuropathy
Acronym: PG-NAION
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FFIS/PG/2017/03
Record Dates: First submitted 2019-01-11; First posted 2019-02-22 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Ischemic Optic Neuropathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alprostadil 20 micrograms (Experimental): 1 μg / kg patient weight up to a maximum of 60 μg
  Interventions: Drug: Alprostadil 20 micrograms
- Placebo (physiological saline solution) (Placebo Comparator): Placebo (physiological saline solution)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Alprostadil 20 micrograms — Intravenous infusion of PGE1 (Days 0, +1 and +2)
  Arms: Alprostadil 20 micrograms
Drug: Placebo — Intravenous infusion of physiological saline solution
  Arms: Placebo (physiological saline solution)

SUMMARY:
Correction of the deficit in the perfusion pressure of the microcirculation that supplies the nerve by intravenous infusion of Prostaglandin E1 (PGE1) (Alprostadil), expected to improve visual function in patients with ischemic optic neuropathy previous non-arteritic (NOIANA).

ELIGIBILITY:
Inclusion criteria:

* Patients of both sexes between the ages of 50 and 80, both inclusive. Patients with the first episode of ischemic optic neuropathy previous non-arteritic / NOIANA. Patients with NOIANA with an evolution time from the beginning of the clinic less than or equal to 15 days.
* Potentially fertile patients should have a negative pregnancy test in serum (beta-HCG / human chorionic gonadotropin) or urine.
* Patients who offer sufficient guarantees of adherence to the protocol.
* Patients who give written informed consent to participate in the study.

Exclusion Criteria:

* Patients with previous optic of any etiology in the affected eye.
* Patients with previous diagnosis or symptoms at the time of arteritis of the temporal artery.
* Patients with optic neuropathy with bilateral clinical presentation of any etiology.
* Patients with loss of vision due to acute hypotension in the context of a surgical intervention, acute hemorrhage or hemodynamic shock.
* Patients with severe loss of previous vision in the eye affected by ophthalmologic causes: severe cataract, glaucoma or intraocular pressure greater than 30 millimeters of mercury, severe diabetic retinopathy, macular degeneration associated with severe age.
* Patients with clinical onset in the month following major non-ocular or intraocular surgery
* Patients with abnormal elevation of CRP / C-reactive protein (> 2 times the upper limit of normal)
* Patients with creatinine levels above 1.5 mg / dL.
* Patients on steroid treatment in the month prior to the episode.
* Patients under treatment with oral anticoagulants.
* Patients on treatment with hydroxychloroquine, ethambutol, vigabatrin at any time before the episode.
* Patients in whom the use of PGE1 (Alprostadil) is contraindicated:
* Patients with participation in a clinical trial in the last 6 months.
* Patients with inability to understand informed consent.
* Pregnant patients, in the postpartum period or during the active lactation period.
* Physically fertile patients

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-06-13 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
determination of visual acuity | Change from baseline visual acuity at 90 days.
  Test ETDRS (Early Treatment Diabetic Retinopathy Study)

SECONDARY OUTCOMES:
Number of Serious Adverse Events | Day 1, day +4,day+30 , day +90.
  Adverse Event
Intraocular Pressure | Day1,day+30 , day +90.
  Intraocular Pressure
Visual Field | Day1,day+30 , day +90.
  Humphrey Field Analyzer (HFA),
Thickness of the layer of nerve fibers and ganglion cells in the retina | Day1,day+30 , day +90.
  Cirrus , Carl Zeiss Meditec, Dublin, California, ver: 6.0.2.81:
fundoscopic evaluation | Day1,day+30 , day +90.
  Biomicroscopy
Hemodynamic indices of the ocular arteries | Day1,day+30 , day +90.
  Doppler SIEMENS Antares™ System:
Optical disc area and cup / disc | Day1,day+30 , day +90.
  Cirrus , Carl Zeiss Meditec, Dublin, California, ver: 6.0.2.81:

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No